CLINICAL TRIAL: NCT01710137
Title: A Placebo Controlled Trial of Varenicline for Smoking Among Those With HIV/AIDS
Brief Title: Varenicline for Nicotine Dependence Among Those With HIV/AIDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01DA033681-01 (NIH); 815435 (Other: University of Pennsylvania Institutional Review Board); R01DA033681 (NIH)
Record Dates: First submitted 2012-10-08; First posted 2012-10-18 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Nicotine Dependence
Keywords: Smoking cessation; Nicotine dependence; Varenicline; Chantix; HIV; AIDS
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Acquired Immunodeficiency Syndrome | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Active Comparator): 12 weeks of active varenicline + smoking cessation counseling
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Interventions: Drug: Varenicline; Behavioral: Smoking Cessation Counseling
- Placebo (Placebo Comparator): 12 weeks of placebo + smoking cessation counseling
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Interventions: Drug: Placebo; Behavioral: Smoking Cessation Counseling

INTERVENTIONS:
Drug: Varenicline
  Other Names: Chantix
  Arms: Varenicline
Drug: Placebo
  Arms: Placebo
Behavioral: Smoking Cessation Counseling

SUMMARY:
Among people diagnosed with HIV/AIDS, the widespread use of highly active antiretroviral therapy (HAART) has greatly improved survival rates and changed the leading causes of death, from AIDS-related diseases to cardiovascular disease and lung cancer. Rates of tobacco use among individuals with HIV/AIDS are very high and varenicline may be particularly efficacious for treating nicotine dependence among individuals with HIV/AIDS. Through this trial, 310 smokers with HIV/AIDS will be randomized to varenicline plus 9 weeks of smoking cessation counseling or placebo plus 9 weeks of smoking cessation counseling. The investigators hypothesize that 1) varenicline and counseling will significantly increase end-of-treatment (week 12) and 24-week biochemically-confirmed abstinence, versus placebo and counseling; 2) quality of life will be rated higher in the varenicline and counseling group versus the placebo and counseling group, and there will be no significant differences between treatment arms in terms of the frequency of severe varenicline-related side effects; and 3) improved affect and reduced cognitive impairment will mediate the effect of varenicline therapy on quit rates.

DETAILED DESCRIPTION:
Among people diagnosed with HIV/AIDS, the widespread use of highly active antiretroviral therapy (HAART) has greatly improved survival rates and changed the leading causes of death, from AIDS-related diseases (e.g., non-Hodgkin's lymphoma, Kaposi sarcoma), to cardiovascular disease and lung cancer. As such, addressing modifiable risk factors for disease mortality among those with HIV/AIDS, including tobacco use, has become a critical priority. To date, only three smoking cessation clinical trials have been conducted with those with HIV/AIDS none of which investigated the efficacy of FDA-approved medications for nicotine dependence. Varenicline is an α4β2 nicotinic acetylcholine receptor partial agonist with greater efficacy for treating nicotine dependence than bupropion or nicotine patch. Varenicline may be particularly efficacious for treating nicotine dependence among individuals with HIV/AIDS given that depression symptoms and cognitive impairment are common in this population, increase during smoking abstinence and predict smoking relapse, and are significantly reduced by varenicline. Therefore, the investigators will conduct a randomized, double-blind, placebo-controlled trial of varenicline with smokers with HIV/AIDS. Specifically, 310 smokers with HIV/AIDS will be randomized to varenicline plus 9 weeks of smoking cessation counseling or placebo plus 9 weeks of smoking cessation counseling. The primary outcome variable for this study will be 7-day biochemically confirmed tobacco abstinence at weeks 12 and 24. Secondary outcomes include: prolonged abstinence to week 12, 18, and 24 (relapse defined as 7 consecutive days of self-reported smoking, after a 2-week grace period), continuous abstinence at weeks 12 and 24 (e.g., no smoking between quit day and follow-up), time to 7-day relapse (no grace period), and lapse and recovery events. The trial results may support the use of varenicline for the treatment of nicotine dependence among those with HIV/AIDS, thereby reducing tobacco-related morbidity and mortality in this population.

ELIGIBILITY:
Inclusion Criteria

1. 18 years of age or older who self-report smoking at least 5 cigarettes (menthol and non-menthol) per day, on average.
2. Diagnosed with HIV infection and exhibiting viral load of < 1000 copies/mL and CD4+ counts of > 200 cells/mm3 within 6 months prior to enrollment.
3. Able to use varenicline safely, based on a medical evaluation including medical history and physical examination, and psychiatric evaluation.
4. Residing in the geographic area for at least 7 months.
5. Women of childbearing potential (based on medical history and physical exam) must consent to use a medically accepted method of birth control (e.g., condoms and spermicide, oral contraceptive, Depo-Provera injection, contraceptive patch, tubal ligation) or abstain from sexual intercourse during the time they are taking study medication and for at least one month after the medication period ends.
6. If current or past diagnosis of bipolar disorder (I, II, or NOS), eligible if:

   1. No psychotic features
   2. MADRS: total score < 8 (past 4 weeks), suicidal item score < 1 (past 4 weeks)
   3. Y-MRS: total score < 8 (past 4 weeks), irritability, speech content, disruptive, or aggressive behavior items score < 3 (past 4 weeks)
   4. No psychiatric hospitalization or Emergency Room visits for psychiatric issues in the past 6 months
   5. No aggressive or violent acts or behavior in the past 6 months
7. Able to communicate fluently in English.
8. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent/HIPAA form.

Exclusion Criteria:

Smoking Behavior

1. Current enrollment or plans to enroll in another smoking cessation program in the next 7 months.
2. Regular (daily) use of chewing tobacco, snuff, snus, cigars, cigarillos, or pipes.
3. Current use or plans to use nicotine substitutes (gum, patch, lozenge, e-cigarette) or smoking cessation treatments in the next 7 months.

   1. Note: Once participants are found eligible for the study, they are told they should refrain from using any nicotine replacement therapy (NRT) for the duration of the study. If a subject reports an isolated (non-daily) instance of NRT use during the study, they may be permitted to continue.

Alcohol/Drug Exclusion Criteria

1. Current untreated and unstable diagnosis of substance abuse or dependence (eligible if past use and if receiving treatment and stable for >30 days).
2. Positive urine drug screen (for cocaine and/or methamphetamines) at the Intake Session.
3. Breath Alcohol Concentration (BrAC) assessment greater than or equal to 0.01 at the Intake Session.

Medication Exclusion Criteria

Current use or recent discontinuation (within last 14 days) of the following medications:

1. Other smoking cessation medications (e.g. Zyban, Wellbutrin, Wellbutrin SR, Chantix)

   a. Note: Once participants are found eligible for the study, they are instructed to only use the smoking cessation medication provided to them by the study staff. If a subject reports an isolated (non-daily) instance of using a non-study smoking cessation medication, the study physician and PI will evaluate the situation and determine if it is safe for the subject to continue participation.
2. Anti-psychotic medications.

Medical Exclusion Criteria

1. Women who are pregnant, planning a pregnancy within the next 7 months, or lactating.
2. Current diagnosis of unstable and untreated major depression, as determined by self-report & MINI (eligible if stable for >30 days).
3. Current or past diagnosis of psychotic disorder, as determined by self-report or MINI.
4. Any suicide risk score on MINI, current suicidal ideation on Columbia scale, or self-reported lifetime suicide attempt.
5. History of heart disease, stroke or MI, unstable angina, or tachycardia (if stable, requires Study Physician approval).
6. Uncontrolled hypertension (SBP >160 or DBP >100).

   a. Note: If a participant presents with blood pressure greater than 160/100 at sessions occurring on Week 0 (Pre-Quit) or at any other point during the treatment period, they will not be provided with/able to continue on medication unless the study physician grants approval.
7. History of kidney or liver failure.
8. Abnormal ECG (unless approved by study physician).
9. Estimated creatinine clearance <50 mL/min, within 6 months prior to enrollment.
10. AST and/or ALT results greater than 2 times the upper limit of normal, within 6 months prior to enrollment.
11. Any impairment (physical, neurological, visual) preventing cognitive task performance.
12. Previous allergic reaction to varenicline.

General Exclusion Criteria

1. Any medical condition or concomitant medication that could compromise subject safety or treatment, as determined by the Principal Investigator and/or Study Physician.
2. Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator and/or Study Physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2012-10; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Schnoll, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Ashare RL, Thompson M, Leone F, Metzger D, Gross R, Mounzer K, Tyndale RF, Lerman C, Mahoney MC, Cinciripini P, George TP, Collman RG, Schnoll R. Differences in the rate of nicotine metabolism among smokers with and without HIV. AIDS. 2019 May 1;33(6):1083-1088. doi: 10.1097/QAD.0000000000002127. PMID 30946162

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline: 12 weeks of active varenicline + smoking cessation counseling
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Varenicline
  Smoking Cessation Counseling
- Placebo: 12 weeks of placebo + smoking cessation counseling
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Placebo
  Smoking Cessation Counseling
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 89 | 90
Completed | 65 | 76
Not Completed | 24 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 89 | 90 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (10.1) | 48.5 (9.7) | 48.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 32 | 57
  Male | 64 | 58 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 9 | 15
  Not Hispanic or Latino | 83 | 81 | 164
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 71 | 72 | 143
  White | 16 | 14 | 30
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 89 | 90 | 179
Time to First Cigarette (TTFC) [Count of Participants; unit: Participants] — Time to first cigarette after waking
  Participants
    Within 5 minutes | 11 | 3 | 14
    6-30 minutes | 3 | 12 | 15
    31-60 minutes | 38 | 38 | 76
    More than 60 minutes | 37 | 37 | 74
Cigarettes/Day in Past 7 Days [Mean (Standard Deviation); unit: Cigarettes] | 11.2 (6.6) | 11.8 (9) | 11.5 (7.9)
Breath CO [Mean (Standard Deviation); unit: ppm] | 15 (10.4) | 13.1 (7.9) | 14.1 (9.2)
Number of Years Smoking [Mean (Standard Deviation); unit: years] | 31.8 (10.8) | 31.1 (11) | 31.5 (10.9)
Number of Times Quit Smoking for>24 Hours [Mean (Standard Deviation); unit: number of times quit smoking] | 8.8 (52.9) | 4.9 (12.3) | 6.9 (38.2)

OUTCOME MEASURES:

1. Primary Outcome: Point Prevalence Tobacco Abstinence
Description: 7-day biochemically-confirmed tobacco abstinence; biochemically-confirmed with urine cotinine.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 89 | 90
Participants | 25 | 11

2. Primary Outcome: Point Prevalence Tobacco Abstinence
Description: 7-day biochemically-confirmed tobacco abstinence; biochemically-confirmed with urine cotinine.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 89 | 90
Participants | 13 | 9

3. Secondary Outcome: Quality of Life at Week 12
Description: The HIV/AIDS-Targeted Quality of Life scale measures overall functioning. Scale range from 7 - 35. Higher score indicates worse quality of life.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 89 | 90
score on a scale | 26.83 (4.49) | 25.95 (4.01)

4. Secondary Outcome: Continuous Abstinence to Week 12
Description: No smoking between the quit day and the follow-up (week 12).
Time Frame: Weeks 12
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 89 | 90
Participants | 21 | 9

5. Secondary Outcome: Continuous Abstinence to Week 24
Description: No smoking between the quit day and the follow-up (Week 24).
Time Frame: Weeks 24
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 89 | 90
Participants | 9 | 6

6. Secondary Outcome: Time to 7-day Relapse
Description: days to smoking regularly for 7 days
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 89 | 90
days | 58.86 (73.90) | 32.48 (62.34)

7. Secondary Outcome: Point Prevalence Tobacco Abstinence
Description: 7-day biochemically-confirmed tobacco abstinence; biochemically-confirmed with urine cotinine.
Time Frame: Week 18
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 89 | 90
Participants | 19 | 10

ADVERSE EVENTS:
Time Frame: 27 weeks
Description: Research staff member completed side effect assessments and determined the severity of the adverse events; the relationship of the event to the study drug and the decision on the course of action for the participant was decided by the site physicians and psychologists after review of the report. Participants were monitored for the development of adverse events by assessing side effects at each assessment time-point, as well as through open-ended questions during assessments.
Arm/Group | Varenicline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/89 | 1/90
Serious Adverse Events (participants affected / at risk) | 5/89 | 3/90
Other Adverse Events (participants affected / at risk) | 19/89 | 28/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=89) | Placebo (N=90)
Death (General disorders) | 0 (0) | 1 (1)
Cancer metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer diagnosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Suicidality (Psychiatric disorders) | 1 (1) | 1 (1)
Hospitalization (General disorders) | 5 (5) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=89) | Placebo (N=90)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dizziness (General disorders) | 1 (1) | 0 (0)
Skin redness (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Weakness (General disorders) | 1 (1) | 0 (0)
ER visit (General disorders) | 0 (0) | 2 (2)
Headache (General disorders) | 3 (3) | 1 (1)
Irritability (General disorders) | 0 (0) | 2 (2)
Hostility (General disorders) | 2 (2) | 5 (5)
Agitation (General disorders) | 8 (8) | 16 (16)
Depression (Psychiatric disorders) | 7 (7) | 16 (16)
Skin swelling (Skin and subcutaneous tissue disorders) | 19 (19) | 28 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT01710137/Prot_SAP_000.pdf